CLINICAL TRIAL: NCT00219778
Title: A Placebo Controlled Study on the Efficacy of 10 mg Oral Mifepristone for the Treatment of Symptomatic Uterine Leiomyomas
Brief Title: A Study on the Efficacy of 10 mg Oral Mifepristone for the Treatment of Symptomatic Uterine Leiomyomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RUFIB
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2010-03

CONDITIONS: Leiomyoma
MeSH Terms: conditions — Leiomyoma | interventions — Mifepristone

INTERVENTIONS:
Drug: mifepristone

SUMMARY:
The first indication of hysterectomies in France are uterine leiomyomas. When they are symptomatic leiomyomas are particularly responsables of an increase of menstruations duration and volume. Echography is the reference exam for the diagnosis. It exists two treatments ways:-firstly progestatives and antifibrinolytics for the treatment of hemorragic symptoms, -secondly LH-RH analogs for the treatment of leiomyomas volume and hemorragic symptoms but just used for a small period because of the risk of osteoporosis.

Different studies with different doses of mifepristone were released. The authors observe a decrease of leiomyomas volume. Based on this experience the present placebo controlled study has for objectives:-to confirm the efficacy of 10 mg oral mifepristone during 24 weeks in the volume decrease and in symptoms of leiomyomas, - to assess the safety of the treatment. The aim is to avoid or delay the hysterectomy of non menopausal patients. During the study patients will be evaluated with biological exams, clinical exams, echographies, medical interrogations and their diary cards.

ELIGIBILITY:
Inclusion Criteria:

* patients who are willing and able to participate in the study
* patients from whom written informed consent has been obtained
* patients who contribute to the National Insurance Scheme
* patients with an age between 25 and 49 years old
* non menopausal patients
* patients who use a non hormonal contraception
* patients with one or several , interstitial or subserous, uterine leiomyomas
* echographic diameter of leiomyomas must be equal or higher than 30 mm
* leiomyomas must be symptomatic

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-12; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of 10 mg oral mifepristone during 24 weeks in the volume decrease of symptomatic uterine leiomymomas

SECONDARY OUTCOMES:
-To determine the efficacy of 10 mg oral mifepristone in symptoms of non menopausal patients with uterine leiomyomas
-To determine the safety of oral mifepristone at the dose of 10 mg per day during 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Magnin, Professor, Principal Investigator — Poitiers University Hospital
Locations (1):
- Poitiers University Hospital, Poitiers, France